CLINICAL TRIAL: NCT04318132
Title: Agreement and Precision Study of the Nidek Mirante OCT Compared to the Optovue RTVue XR Avanti OCT and SLO Image Comparison of the Nidek Mirante and the OPTOS P200DTx
Brief Title: Agreement and Precision Study of the Nidek Mirante
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Nidek Mirante-001
Record Dates: First submitted 2020-02-12; First posted 2020-03-23 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Glaucoma; Retinal Disease; Corneal Disease
MeSH Terms: conditions — Glaucoma; Retinal Diseases; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- NIDEK Mirante Comparison - Normal (Experimental): Subjects without any current ocular pathology other than cataract in either eye
  Interventions: Device: Nidek Mirante; Device: Optovue RTVue XR Avanti; Device: Optos P200DTx
- NIDEK Mirante Comparison - Retina (Experimental): Subjects diagnosed with retinal pathology
  Interventions: Device: Nidek Mirante; Device: Optovue RTVue XR Avanti; Device: Optos P200DTx
- NIDEK Mirante Comparison - Glaucoma (Experimental): Subjects who have been diagnosed with glaucoma
  Interventions: Device: Nidek Mirante; Device: Optovue RTVue XR Avanti; Device: Optos P200DTx
- NIDEK Mirante Comparison - Corneal disease (Experimental): Subjects with corneal pathologies
  Interventions: Device: Nidek Mirante; Device: Optovue RTVue XR Avanti

INTERVENTIONS:
Device: Nidek Mirante — The Nidek Mirante Optical Coherence Tomography (OCT) including scanning laser ophthalmoscope (SLO) function is an non-contact system for imaging the fundus and for axial cross sectional imaging of anterior and posterior ocular structures.
Device: Optovue RTVue XR Avanti — The Avanti is an optical coherence tomography system indicated for the in vivo imaging,axial cross-sectional, and three-dimensional imaging and measurement of anterior and posterior ocular structures.
Device: Optos P200DTx — The P200DTx scanning laser ophthalmoscope (SLO) is indicated for use as a widefield and retinal fluorescence and autofluorescence imaging ophthalmoscope to aid in the diagnosis and monitoring of diseases and disorders that manifest in the retina.
  Arms: NIDEK Mirante Comparison - Glaucoma; NIDEK Mirante Comparison - Normal; NIDEK Mirante Comparison - Retina

SUMMARY:
This study is a prospective comparative, randomized, single center study to gather agreement and precision of the Nidek Mirante OCT with SLO and Anterior Segment Imaging capabilities in comparison to the Optovue RTVue XR Avanti OCT and Optos P200DTx in normal subjects, subjects with glaucoma, subjects with retinal disease and subjects with corneal disease.

DETAILED DESCRIPTION:
This is a prospective comparative clinical study to be conducted at one clinical site located in the United States. Three Nidek Mirante devices, three Optovue RTVue XR Avanti devices and one OPTOS P200DTx will be used. For agreement and precision analysis of OCT scans and agreement analysis of image quality of OCT ACA scans, each Nidek Mirante device will be paired with one of the Optovue RTVue XR Avanti devices. One device operator will be assigned to each device pair to create three distinct operator/device configurations.

For agreement analysis of SLO image quality, one OPTOS P200DTx will be included in one of three operator/device configurations.

ELIGIBILITY:
Inclusion Criteria - Normal Group:

1. Male or female subjects from 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects with normal eye examinations (without pathology other than cataract) in both eyes on the date of the study visit as observed with a +90 Diopter Fundus Lens;
5. Subjects with current best-spectacle-corrected visual acuity (BSCVA) of 20/40 or better in both eyes on the date the study visit.

Exclusion Criteria - Normal Group:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in either eye;
3. Subjects with any current ocular pathology other than cataract in either eye, as determined by self-report and confirmed by the investigator assessment and/or confirmed by the investigator assessment at the study visit;
4. Subjects with (or history of) leukemia, dementia or multiple sclerosis;
5. Subject has a condition or will be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Inclusion Criteria - Glaucoma Group:

1. Male or female subjects from 22 years of age or older who have full legal capacity to volunteer on the date the informed consent was signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects who have been diagnosed with glaucoma in the glaucoma study eye(s), with optic nerve damage as evidenced by either of the following optic disc or RNFL structural abnormalities observed via fundus exam during the study visit:

   1. Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage; or
   2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue;
5. Subjects with a current BSCVA of 20/40 or better in the glaucoma study eye(s) on the date of the visit;
6. History of a reliable Humphrey Field Analyzer (HFA) visual field (24-2 SITA Standard, white on white) measured on the day of study visit 1, or within the previous six (6) months from study visit 1 with reliable results, defined as fixation losses < 20%, or false positives < 33%, or false negatives < 33% in the glaucoma study eye(s) that is consistent with glaucomatous optic nerve damage in glaucoma study eye(s) based on at least one of the following findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level; or
   2. Glaucoma hemi-field test "outside normal limits."

Exclusion Criteria - Glaucoma Group:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in the glaucoma study eye(s);
3. Subjects with retinal disease in the glaucoma study eye(s), as determined by self-report and confirmed by the investigator assessment and/or confirmed by the investigator assessment at the study visit;
4. Subjects with (or history of) leukemia, dementia or multiple sclerosis;
5. Subject has a condition or will be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Inclusion Criteria - Retinal Disease Group:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects with a current BSCVA of 20/400 or better in the retinal disease study eye(s) at the study visit;
5. Subjects diagnosed with retinal pathology including but not limited to: Non Exudative Macular Degeneration (dry AMD), Diabetic Macular Edema, Macular Hole, Epiretinal Membrane, Cystoid Macular Edema, or other retinal disease in the study eye(s) as confirmed within the past six (6) months, who exhibit structural lesions in the study eye.

Exclusion Criteria - Retinal Disease Group

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in the study eye;
3. Subjects with glaucoma in the retinal disease study eye(s), as determined by self-report and confirmed by the investigator assessment and/or confirmed by the investigator assessment at the study visit;
4. Subjects with (or history of) leukemia, dementia or multiple sclerosis;
5. Subject has a condition or will be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Inclusion Criteria - Corneal Group

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects with a current BSCVA of 20/400 or better in the study eye(s) at the study visit;
5. Subjects with corneal pathologies including but not limited to: Post status LASIK surgery, Keratoconus, or other corneal dystrophies or degenerations in the study eye(s) as confirmed within the past six (6) months.

Exclusion Criteria - Corneal Group

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images in the study eye;
3. Subjects with (or history of) leukemia, dementia or multiple sclerosis;
4. Subject has a condition or will be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tadakazu Ichimura, Study Director — Nidek Co. LTD.
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- NIDEK Mirante Comparison - Corneal Disease: Subjects who have been diagnosed with corneal pathologies
Period: Overall Study
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Retina | NIDEK Mirante Comparison - Glaucoma | NIDEK Mirante Comparison - Corneal Disease
Started | 45; 45 eyes | 47; 47 eyes | 46; 46 eyes | 32; 32 eyes
Completed | 45; 45 eyes | 47; 47 eyes | 43; 43 eyes | 32; 32 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes | 3; 3 eyes | 0; 0 eyes
Not completed — Protocol Violation | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Retina | NIDEK Mirante Comparison - Glaucoma | NIDEK Mirante Comparison - Corneal Disease | Total
Number analyzed (Participants) | 45 | 47 | 46 | 32 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 16 | 18 | 21 | 96
  >=65 years | 4 | 31 | 28 | 11 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (15.36) | 69.7 (11.23) | 65.1 (9.20) | 55.4 (15.09) | 59.2 (16.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 25 | 20 | 99
  Male | 17 | 21 | 21 | 12 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 1 | 5
  White | 41 | 46 | 42 | 29 | 158
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 47 | 46 | 32 | 170

OUTCOME MEASURES:

1. Primary Outcome: Agreement of Macular Thickness (μm) Measurement for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Agreement of the measured Macular thickness (μm) between the test device and the predicate device for the OCT function of NIDEK Mirante.
Time Frame: 1 day
Population: The cornea arm/group was omitted because this group did not measure the macular thickness.
Measure: Mean (Standard Deviation); unit: μm
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Retina | NIDEK Mirante Comparison - Glaucoma
Number analyzed (Participants) | 45 | 46 | 43
Number analyzed (eyes) | 45 | 46 | 43
μm
  Center | 10.658 (4.3789) | 11.032 (6.9749) | 11.415 (4.8615)
  Inner Temporal | 19.200 (6.4194) | 17.065 (4.2079) | 17.047 (6.2104)
  Inner Superior | 22.889 (6.0386) | 18.870 (3.8965) | 20.628 (5.8879)
  Inner Nasal | 21.911 (6.0521) | 19.043 (4.5896) | 19.721 (6.1965)
  Inner Inferior | 22.267 (4.7645) | 19.739 (5.4014) | 19.163 (7.3870)
  Outer Temporal | 10.267 (6.5796) | 9.587 (5.2560) | 9.628 (5.3275)
  Outer Superior | 11.311 (5.4306) | 10.370 (6.0309) | 10.767 (6.2786)
  Outer Nasal | 12.733 (6.0317) | 10.522 (6.4524) | 11.023 (5.8614)
  Outer Inferior | 13.844 (5.5757) | 11.957 (7.4951) | 12.581 (6.3555)

2. Primary Outcome: Agreement of Retinal Nerve Fiber Layer Thickness (μm) Measurement for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Agreement of the measured Retinal nerve fiber layer thickness around Optic nerve head between the test device and the predicate device for the OCT function of NIDEK Mirante.
Time Frame: 1 day
Population: The retina and cornea arm/group were omitted because this group did not measure the retinal nerve fiber layer thickness.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Glaucoma
Number analyzed (Participants) | 45 | 43
Number analyzed (eyes) | 45 | 43
µm
  Whole Chart | 9.233 (4.3936) | 7.536 (4.7895)
  S/I Inferior | 9.725 (5.3925) | 7.631 (7.0398)
  S/I Superior | 8.554 (5.5885) | 7.426 (7.1255)
  TSNIT Temporal | -4.515 (8.1383) | 1.965 (10.0886)
  TSNIT Superior | 11.762 (8.8701) | 5.928 (10.1354)
  TSNIT Nasal | 12.250 (8.7671) | 12.395 (7.7614)
  TSNIT Inferior | 17.211 (8.6067) | 9.854 (8.5394)
  Horizontal C/D Ratio | 0.018 (0.1977) | -0.061 (0.1358)
  Vertical C/D Ratio | 0.030 (0.1944) | -0.056 (0.1401)
  Disc Area | 0.271 (0.1995) | 0.210 (0.2919)
  Cup Area | 0.055 (0.2236) | -0.010 (0.2491)

3. Primary Outcome: Agreement of Corneal Thickness (μm) Measurement for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Agreement of the measured Corneal thickness between the test device and the predicate device for the OCT function of NIDEK Mirante.
Time Frame: 1 day
Population: The retina and glaucoma arm/group were omitted because this group did not measure the corneal thickness.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Corneal Disease
Number analyzed (Participants) | 45 | 19
Number analyzed (eyes) | 45 | 19
µm | 16.511 (3.9117) | 14.842 (8.3084)

4. Primary Outcome: Agreement of SLO Image Quality (Likert Scale) for Nidek Mirante and OPTOS P200DTx
Description: Agreement of the SLO Image quality between the test device and the predicate device for the SLO function of NIDEK Mirante.
  The image quality of is graded Clinical Utility and Overall Utility for each image patterns (SLO Color Fundus, SLO B-FAF and SLO G-FAF) on a Likert scale. The grading used the 0-3 point scale, and higher scores mean a better image quality.
Time Frame: 1 day
Population: Some patients could not be captured acceptable SLO images. The cornea arm/group was omitted because this group was not included in the SLO images assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Retina | NIDEK Mirante Comparison - Glaucoma
Number analyzed (Participants) | 45 | 47 | 43
Number analyzed (eyes) | 45 | 47 | 43
score on a scale
  SLO Color Fundus: Clinical Utility: number analyzed (Participants) | 44 | 47 | 36
  SLO Color Fundus: Clinical Utility | 2.9 (0.21) | 2.9 (0.27) | 3.0 (0.11)
  SLO Color Fundus: Overall Quality: number analyzed (Participants) | 44 | 47 | 36
  SLO Color Fundus: Overall Quality | 3.0 (0.17) | 2.8 (0.37) | 3.0 (0.11)
  SLO B-FAF: Clinical Utility: number analyzed (Participants) | 42 | 46 | 34
  SLO B-FAF: Clinical Utility | 2.6 (0.48) | 2.3 (0.62) | 2.6 (0.41)
  SLO B-FAF: Overall Quality: number analyzed (Participants) | 42 | 46 | 34
  SLO B-FAF: Overall Quality | 2.6 (0.52) | 2.2 (0.67) | 2.5 (0.49)
  SLO G-FAF: Clinical Utility: number analyzed (Participants) | 42 | 47 | 35
  SLO G-FAF: Clinical Utility | 2.4 (0.61) | 2.4 (0.53) | 2.6 (0.41)
  SLO G-FAF: Overall Quality: number analyzed (Participants) | 42 | 47 | 35
  SLO G-FAF: Overall Quality | 2.4 (0.65) | 2.4 (0.54) | 2.6 (0.47)

5. Primary Outcome: Agreement of the ACA Image Quality (Likert Scale) for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Agreement of the ACA Image quality between the test device and the predicate device for the OCT function of NIDEK Mirante.
  The image quality of is graded Clinical Utility and Overall Utility on a Likert scale. The grading used the 0-3 point scale, and higher scores mean a better image quality.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Retina | NIDEK Mirante Comparison - Glaucoma | NIDEK Mirante Comparison - Corneal Disease
Number analyzed (Participants) | 44 | 46 | 42 | 32
Number analyzed (eyes) | 44 | 46 | 42 | 32
score on a scale
  Clinical Utility | 2.4 (0.39) | 2.2 (0.42) | 2.3 (0.43) | 2.2 (0.56)
  Overall Utility | 2.2 (0.47) | 2.1 (0.45) | 2.2 (0.45) | 2.1 (0.54)

6. Primary Outcome: Precision of the Macular Thickness (μm) Measurement for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Precision (repeatability) of the measured Full retinal thickness at Macula for the OCT function of the NIDEK TONOREF III.
Time Frame: 1 day
Population: The cornea arm/group was omitted because this group did not measure the Full retinal thickness at Macula.
Measure: Number; unit: %CV Repeatability
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Retina | NIDEK Mirante Comparison - Glaucoma
Number analyzed (Participants) | 44 | 44 | 40
Number analyzed (eyes) | 44 | 44 | 40
%CV Repeatability
  Center | 1.034 | 1.163 | 1.031
  Inner Temporal | 0.425 | 0.863 | 0.433
  Inner Superior | 0.606 | 0.701 | 0.531
  Inner Nasal | 0.465 | 0.608 | 0.441
  Inner Inferior | 0.502 | 0.806 | 0.678
  Outer Temporal | 0.764 | 0.971 | 0.786
  Outer Superior | 0.682 | 0.776 | 0.784
  Outer Nasal | 0.415 | 0.593 | 0.528
  Outer Inferior | 0.865 | 1.075 | 1.012

7. Primary Outcome: Precision of the Retinal Nerve Fiber Layer Thickness (μm) Measurement for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Precision (repeatability) of the measured Retinal nerve fiber layer thickness around Optic nerve head at Macula for the OCT function of the NIDEK TONOREF III.
Time Frame: 1 day
Population: The retina and cornea arm/group were omitted because these groups did not measure the retinal nerve fiber layer thickness around the Optic nerve head.
Measure: Number; unit: %CV Repeatability
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Glaucoma
Number analyzed (Participants) | 40 | 34
Number analyzed (eyes) | 40 | 34
%CV Repeatability
  TSNIT Inferior | 3.813 | 6.015
  TSNIT Nasal | 6.730 | 7.814
  TSNIT Superior | 3.708 | 6.495
  TSNIT Temporal | 4.514 | 7.703
  Whole Chart | 2.268 | 3.531
  S/I Inferior | 3.950 | 5.563
  S/I Superior | 3.550 | 5.900
  Horizontal C/D Ratio | 9.380 | 6.725
  Vertical C/D Ratio | 7.394 | 5.912
  Disc Area | 5.892 | 7.553
  Cup Area | 14.148 | 10.047

8. Primary Outcome: Precision of the Corneal Thickness (μm) Measurement for Nidek Mirante and Optovue RTVue XR Avanti OCT
Description: Precision (repeatability) of the measured Thickness of the Cornea for the OCT function of the NIDEK TONOREF III.
Time Frame: 1 day
Population: The retina and glaucoma arm/group were omitted because these groups did not measure the thickness of the cornea.
Measure: Number; unit: %CV Repeatability
Units Other Than Participants: eyes
Arm/Group | NIDEK Mirante Comparison - Normal | NIDEK Mirante Comparison - Corneal Disease
Number analyzed (Participants) | 42 | 18
Number analyzed (eyes) | 42 | 18
%CV Repeatability | 0.535 | 0.878

9. Secondary Outcome: Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational device but not necessarily related to the investigational device.
Time Frame: 1 day
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Groups:
- Normals; Retina; Glaucoma: Nidek Mirante: The Nidek Mirante Optical Coherence Tomography (OCT) including scanning laser ophthalmoscope (SLO) function is an non-contact system for imaging the fundus and for axial cross sectional imaging of anterior and posterior ocular structures.
  Optovue RTVue XR Avanti: The Avanti is an optical coherence tomography system indicated for the in vivo imaging,axial cross-sectional, and three-dimensional imaging and measurement of anterior and posterior ocular structures.
  Optos P200DTx: The P200DTx scanning laser ophthalmoscope (SLO) is indicated for use as a widefield and retinal fluorescence and autofluorescence imaging ophthalmoscope to aid in the diagnosis and monitoring of diseases and disorders that manifest in the retina.
- Corneal Disease: Nidek Mirante: The Nidek Mirante Optical Coherence Tomography (OCT) including scanning laser ophthalmoscope (SLO) function is an non-contact system for imaging the fundus and for axial cross sectional imaging of anterior and posterior ocular structures.
  Optovue RTVue XR Avanti: The Avanti is an optical coherence tomography system indicated for the in vivo imaging,axial cross-sectional, and three-dimensional imaging and measurement of anterior and posterior ocular structures.
Arm/Group | Normals | Retina | Glaucoma | Corneal Disease
Number analyzed (Participants) | 45 | 47 | 46 | 32
Number analyzed (eyes) | 45 | 47 | 46 | 32
eyes | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Normals | Retina | Glaucoma | Corneal Disease
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47 | 0/46 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47 | 0/46 | 0/32
Other Adverse Events (participants affected / at risk) | 0/45 | 0/47 | 0/46 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT04318132/Prot_SAP_001.pdf